CLINICAL TRIAL: NCT05087316
Title: Biometric Oral Appliance Therapy for the Treatment of Obstructive Sleep Apnea in Adults
Brief Title: Therapy of Oral Appliance for Adults Jordanians With Obstructive Sleep Apnea
Acronym: TOAAJOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 314/2017
Record Dates: First submitted 2021-09-22; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Mild Obstructive Sleep Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator)
  Interventions: Device: Standard hospital treatment
- Oral Appliance (Experimental)
  Interventions: Device: biomimetic oral appliance therapy (BOAT)

INTERVENTIONS:
Device: biomimetic oral appliance therapy (BOAT) — BOAT appliance is designed to correct maxillo-mandibular underdevelopment in both children and adults (Singh and Lipka, 2009). However, adults will only use for this study. Typically, a BOAT appliance consists of 6 patented, anterior 3-D Axial Springs™, a midline actuator (such as omega loops or screws), posterior occlusal rests, and a round labial bow (Figure 1). Patients will be trained on activation of the screw
  Arms: Oral Appliance
Device: Standard hospital treatment — Use of CPAP and similar methods
  Arms: Standard treatment

SUMMARY:
Introduction: Obstructive Sleep Apnea (OSA) is the most common form of sleep disordered breathing. Patients who arrive at the dental office with a diagnosis of OSA are often treated with a mandibular advancement device (MAD). A biomimetic oral appliance therapy (BOAT), offers an alternative non-surgical method, which can putatively resolve OSA by combined maxilla-mandibular correction, and addressing craniofacial deficiencies.

The aim: To determine whether maxilla-mandibular correction changes induced by BOAT produce a more favorable upper airway, which might result in a reduction in the severity of OSA.

Protocol: Adults who underwent an overnight sleep study and were diagnosed by a sleep specialist physician will be potential subjects for the current study. The BQ and EES will be recorded pre- and post- BOAT treatment. Subjects with mild to moderate OSA will have 2 months follow up visits and a final overnight sleep study to measure apnea-hypopnea index (AHI). The subjects will be asked to wear the appliance for 10-12 hours/day and at night. Findings will be analyzed statistically using paired t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mild to moderate OSA with good oral hygiene
* Intolerant to CPAP therapy
* Having enough number of maxillary and mandibular teeth to retain the removable device.

Exclusion Criteria:

* Patients who are unable to attend regular appointments and unable to consent.
* Patients with severe OSA who met the inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
AHI | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King abdullah University Hospital (KAUH), Irbid, Others, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khasawneh L, Al Mortadi N, Abu-Ishqair E, Khassawneh B, Alzoubi KH. Cone beam computed tomography changes upon oral appliance therapy for adult patients with obstructive sleep apnea: A non-randomized clinical trial. Medicine (Baltimore). 2024 Oct 4;103(40):e39923. doi: 10.1097/MD.0000000000039923. PMID 39465752